CLINICAL TRIAL: NCT07294586
Title: Exploratory Clinical Study and Validation of Blood Biomarkers for Alzheimer's Disease
Acronym: ADKIT
Status: Completed | Type: Observational
Sponsor: Amoneta Diagnostics SAS (Industry)
Collaborators: Hopitaux Civils de Colmar (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-AMDx.001; 2015-A00118-41 (Registry Identifier: RCB)
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-10

CONDITIONS: Alzheimer Disease; Dementia; Neurodegenerative Disorders; Cognitive Decline; Memory Loss; Mild Cognitive Impairment (MCI); Early Onset Alzheimer Disease; Late Onset Alzheimer Disease
Keywords: Alzehimer's Disease; Blood Biomarkers; Protein Kinase C (PKC); Amyloid Beta; Neurodegeneration; Early Diagnosis; AD Patients
MeSH Terms: conditions — Alzheimer Disease; Dementia; Neurodegenerative Diseases; Cognitive Dysfunction; Memory Disorders; Plaque, Amyloid; Nerve Degeneration; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, urine, and RNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 - Healthy volunteers: This group includes cognitively healthy individuals aged 50 to 85 years, with no clinical signs of neurodegenerative disease. Participants will undergo clinical evaluation, routine blood and urine sampling, and neuropsychological testing. Samples will be used to establish baseline biomarker levels and support biobank development.
  Sample Size: 100 participants
- Group 2 - AD patients: This group includes patients aged 50 to 85 years diagnosed with Alzheimer's disease based on clinical criteria, neuropsychological testing, and imaging. Participants will undergo comprehensive clinical evaluation and biological sampling to assess biomarker performance.
  Sample Size: 100 participants

SUMMARY:
This is a 24-month, monocentric, exploratory and observational clinical study aimed at developing and validating a blood-based diagnostic test for Alzheimer's disease (AD). The test is based on two complementary biomarkers: conformational changes in Protein Kinase C (PKC) and aggregation of β-amyloid peptide on red blood cell membranes. The study will also establish a biobank of serum, plasma, urine, and RNA samples for future biomarker research.

ELIGIBILITY:
Inclusion Criteria:

For All Participants (HV and AD groups):

* Age between 50 and 85 years
* Ability to understand and sign informed consent
* Availability for the full duration of the study (24 months)
* Fasting capability for morning sample collection (between 8:30-12:00)
* Willingness to provide blood and urine samples for biomarker analysis and biobank storage

Additional Criteria for Healthy Volunteers (HV):

* No history or current diagnosis of neurodegenerative disease
* Normal cognitive function confirmed by neuropsychological testing (e.g., MMSE score within normal range)
* No significant abnormalities on brain imaging (CT or MRI if performed)
* No use of medications affecting cognitive function

Additional Criteria for Alzheimer's Disease Patients (AD):

* Clinical diagnosis of probable Alzheimer's disease based on standardized criteria
* Cognitive impairment confirmed by neuropsychological testing (e.g., MMSE score below threshold)
* Supporting evidence from brain imaging (CT or MRI) and/or cerebrospinal fluid biomarkers (if available)
* Stable medical condition allowing participation in study procedures

Exclusion Criteria:

For All Participants:

* History of major psychiatric disorders (e.g., schizophrenia, bipolar disorder)
* Significant neurological conditions other than Alzheimer's disease (e.g., Parkinson's disease, stroke)
* Active malignancy or history of cancer within the past 5 years (except localized skin cancer)
* Severe renal, hepatic, or cardiovascular disease
* Current participation in another interventional clinical trial
* Known blood disorders or conditions affecting red blood cell morphology or function
* Recent blood transfusion (within 3 months)
* Substance abuse or alcohol dependence
* Inability to comply with study procedures

Additional Exclusion for Healthy Volunteers:

* Any cognitive complaints or subjective memory loss
* First-degree family history of Alzheimer's disease (optional, depending on stratification strategy)
* Use of psychoactive medications

Additional Exclusion for Alzheimer's Disease Patients:

* Diagnosis of mixed or atypical dementia
* Rapidly progressive cognitive decline suggestive of other pathology
* Contraindications to lumbar puncture (if CSF sampling is planned)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of 200 individuals aged 50 to 85 years, divided into two cohorts:
  Healthy Volunteers (HV): 100 cognitively healthy individuals with no history of neurodegenerative disease. These participants will serve as controls for biomarker comparison.
  Alzheimer's Disease Patients (AD): 100 individuals clinically diagnosed with probable Alzheimer's disease based on neuropsychological testing, clinical evaluation, and imaging. These participants represent the target population for biomarker validation.
  Participants will be stratified by age and sex to ensure balanced representation across both groups. All subjects must be able to provide informed consent and comply with study procedures, including fasting sample collection and clinical assessments.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2021-06-24 (Actual)

PRIMARY OUTCOMES:
Quantification of Blood Biomarkers in Alzheimer's Disease and Healthy Subjects | At baseline (Visit 0)
  Measurement and comparison of two blood-based biomarkers-(1) conformational change in Protein Kinase C (PKC) and (2) aggregation of β-amyloid peptide (Aβ1-42) on red blood cell membranes-between patients diagnosed with Alzheimer's disease and age- and sex-matched healthy volunteers. The goal is to assess the diagnostic performance of each biomarker individually.

SECONDARY OUTCOMES:
Analytical Performance of Biomarkers Across Demographic and Clinical Variables | Within 1 month after sample collection
  Evaluation of the influence of age, sex, sample matrix (serum, plasma, urine), and storage conditions on the analytical performance of each biomarker.
Establishment of a Biobank for Future Biomarker Research | Throughout the 24-month study period
  Collection and storage of biological samples (serum, plasma, urine, RNA) from all participants to support future studies on Alzheimer's disease and related biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: François Sellal, MD, Principal Investigator — Hopitaux Civils de Colmar
Locations (1):
- Hôpitaux Civils de Colmar, Colmar, Alsace, France